CLINICAL TRIAL: NCT03102996
Title: Preservation of Kidney Function in Kidney Transplant Recipients by Alkali Therapy (Preserve-Transplant Study): a Multi-center Randomized Single-blind Placebo- Controlled Trial
Brief Title: Preserve-Transplant Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Preserve-Transplant Study
Record Dates: First submitted 2017-03-31; First posted 2017-04-06 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Acidosis; Renal Insufficiency; Kidney Transplantation
Keywords: Alkali; Graft; Acid base; Metabolic acidosis; Chronic kidney disease
MeSH Terms: conditions — Acidosis; Renal Insufficiency; Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Verum (Experimental): Patients will receive Nephrotrans.
  Interventions: Drug: Nephrotrans
- Placebo (Placebo Comparator): Patients will receive Placebo.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Nephrotrans — Sodium hydrogen carbonate, ATC-Code: A02AH
  Arms: Verum
Other: Placebo — Identical capsules without active substance.
  Arms: Placebo

SUMMARY:
The aim of this study is to test if alkali treatment will preserve kidney graft function and diminish the progression of chronic kidney disease in renal transplant patients. Additionally the underlying mechanisms of nephrotoxicity of metabolic acidosis will be investigated in this cohort.

This study is a multi-center, prospective, randomized, single-blind (patient), placebo-controlled interventional trial to test the superiority of alkali treatment in comparison to placebo on preservation of kidney function in 300 kidney transplant recipients. The duration of the study will be 2 years for the individual participant. The patients will be randomized into 2 arms: intervention arm (sodium hydrogen carbonate, product: Nephrotrans®) and placebo arm (placebo comparator).

Several studies in CKD (chronic kidney disease) patients have shown that alkali therapy slows progression of CKD.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent as documented by signature
* age ≥ 18 years and able to give informed consent
* ≥ 12 months after renal transplantation
* stable clinical condition
* stable graft function over the last 3 months (creatinine changes ± 15%)
* eGFR between 15-89 ml/min/1.73 m2
* serum bicarbonate ≤ 22 mmol/l within the last 6 months

Exclusion Criteria:

* uncontrolled hypertension or use of > 4 antihypertensive agents
* uncontrolled heart failure
* serum potassium < 3.0 mmol/l
* serum sodium > 150 mmol/l
* use of alkali in the preceding 4 weeks
* use of mineralocorticoid antagonists, topiramate, carbo anhydrase inhibitors or any drugs with similar effects
* history of noncompliance with clinic visits
* hereditary fructose intolerance
* known hypersensitivity or allergy to the drug used in this study or to peanut, sorbitol, and soy
* pregnancy or breastfeeding
* intention to become pregnant during the course of the study
* lack of safe contraception, defined as: Female participants of childbearing potential, not using and not willing to continue using a medically reliable method of contraception for the entire study duration, such as oral, injectable, or implantable contraceptives, or intrauterine contraceptive devices, or who are not using any other method considered sufficiently reliable by the investigator in individual cases.
* please note that female participants who are surgically sterilised / hysterectomised or post-menopausal for longer than 2 years are not considered as being of child bearing potential.
* suspected drug or alcohol abuse
* inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant
* enrolment of the investigator, his/her family members, employees and other dependent persons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2017-06-12 (Actual); Primary Completion 2021-06-29 (Actual); Study Completion 2021-07-26 (Actual)

PRIMARY OUTCOMES:
eGFR | 2 years
  Change in renal function by assessing the change in eGFR over 2 years from baseline. eGFR will be determined based on the CKD-EPI creatinine equation.

CONTACTS AND LOCATIONS:
Overall Officials: Nilufar Mohebbi, PD Dr. med., Principal Investigator — University of Zurich; Rudolf P Wüthrich, Prof. Dr. med., Study Director — University of Zurich
Locations (3):
- Switzerland (3):
  - Inselspital Bern, Department of Nephrology and Hypertension, Bern, Canton of Bern
  - HUG - Néphrologie, Geneva, Canton of Geneva
  - University Hospital Zurich, Division of Nephrology, Zurich, Canton of Zurich

REFERENCES:
- [Derived] Mohebbi N, Ritter A, Wiegand A, Graf N, Dahdal S, Sidler D, Arampatzis S, Hadaya K, Mueller TF, Wagner CA, Wuthrich RP. Sodium bicarbonate for kidney transplant recipients with metabolic acidosis in Switzerland: a multicentre, randomised, single-blind, placebo-controlled, phase 3 trial. Lancet. 2023 Feb 18;401(10376):557-567. doi: 10.1016/S0140-6736(22)02606-X. Epub 2023 Jan 25. PMID 36708734
- [Derived] Wiegand A, Ritter A, Graf N, Arampatzis S, Sidler D, Hadaya K, Muller TF, Wagner CA, Wuthrich RP, Mohebbi N. Preservation of kidney function in kidney transplant recipients by alkali therapy (Preserve-Transplant Study): rationale and study protocol. BMC Nephrol. 2018 Jul 13;19(1):177. doi: 10.1186/s12882-018-0956-8. PMID 30001705